CLINICAL TRIAL: NCT00804128
Title: Contrast-enhanced MRI for the Characterization of Ductal Carcinoma in Situ (DCIS)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000616972; 08755 (Other: University of California, San Francisco); NCI-2019-07528 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA116182 (NIH); U01CA225427 (NIH); R01CA249016 (NIH)
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Magnetic Resonance Spectroscopy; gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Cancer patients: Adult, breast cancer patients with confirmed Ductal Carcinoma in Situ (DCIS) or atypical ductal hyperplasia (ADH)
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Drug: Gadavist

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI
  Other Names: MRI
Drug: Gadavist — Gadavist injection is a paramagnetic macrocyclic contrast agent administered for magnetic resonance imaging
  Other Names: Gadobutrol

SUMMARY:
*REFERRALS TO THIS TRIAL MUST BE THROUGH BREAST CARE CLINICIANS ONLY*

RATIONALE: Diagnostic procedures, such as contrast-enhanced MRI, may help find and diagnose ductal carcinoma in situ.

PURPOSE: This study is to develop and refine magnetic resonance (MR) imaging methods for pre-operative staging of ductal carcinoma in situ, a pre-invasive form of breast cancer, and atypical ductal hyperplasia, a risk factor for developing cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the DCIS optimized MRI to the standard clinical MRI. Using a scale of 1-5 from poor to excellent, images will be assessed for conspicuity of DCIS and atypical ductal hyperplasia (ADH) lesions, agreement of disease extent with biopsy, and overall image quality (artifact level, uniformity of fat suppression, contrast to noise ratio and signal to noise ratio).
* Subjects with ADH, a benign condition that can also show enhancement on MRI, will be enrolled to explore the utility of the DCIS optimized MRI for distinguishing DCIS and ADH.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patients at the University of California, San Francisco Breast Care Center meeting the following criteria:

    * Biopsy proven ductal carcinoma in situ (DCIS) of the breast.
    * Has undergone mammography within the past 60 days.
    * ADH patients: over 18, no prior history of breast disease.

PATIENT CHARACTERISTICS:

* Referrals to this trial are through breast care clinicians only
* Not pregnant or nursing (or stopped nursing within the past 3 months)
* Negative pregnancy test
* No contraindication to MRI (e.g., implanted pacemaker, implanted ferromagnetic device, ferromagnetic aneurysm clip, severe claustrophobia, ocular metal fragments, or shrapnel injury)

PRIOR CONCURRENT THERAPY:

* More than 2 years since prior surgery to the ipsilateral breast (patient)
* No prior radiotherapy to the ipsilateral breast (patient)
* No prior cytotoxic regimens (patient)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving care for breast cancer who also have a biopsy proven DCIS or ADH.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Comparison of ductal carcinoma in situ (DCIS)-optimized MRI quality | 1 month
  Conspicuity of DCIS lesion, agreement of disease extent with biopsy, and overall image quality will be used to determine the overall image quality for each MRI.
Comparison of two DCIS-optimized MRIs for variability in enhancement levels for DCIS | 1 month
  Conspicuity of DCIS lesion, agreement of disease extent with biopsy, and overall image quality will be used to determine the overall image variability for each MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Nola M. Hylton, PhD, Principal Investigator — University of California, San Francisco; Bonnie Joe, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT00804128/ICF_000.pdf